CLINICAL TRIAL: NCT03298022
Title: Efficacy and Safety of ALTB-168 in Patients With Moderate to Severe Active, Anti-TNF Alpha and/or Anti-integrin Refractory Ulcerative Colitis: a 26-week, Open-label, Multi-center, Phase II Proof of Principle Trial
Brief Title: Efficacy&Safety of ALTB-168 in Patients With Moderate to Severe Active,Anti-TNF Alpha and/or Anti-integrin Refractory UC
Acronym: TNF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: As a consequence of operational difficulties at the clinical sites associated with the COVID-19 pandemic
Sponsor: AltruBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017.008.01
Record Dates: First submitted 2017-09-27; First posted 2017-09-29 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALTB-168 (Experimental): intravenous doses of ALTB-168
  Interventions: Biological: ALTB-168

INTERVENTIONS:
Biological: ALTB-168 — monoclonal antibody
  Other Names: Neihulizumab

SUMMARY:
To evaluate the efficacy and safety of Neihulizumab (ALTB-168) administered intravenously in patients with moderate to severe active ulcerative colitis who are refractory or intolerant to anti-Tumor Necrosis Factor α and/or anti-integrin treatments.

DETAILED DESCRIPTION:
This is a Phase II, open label, single arm, multiple dose proof of principle study to test the efficacy and safety of Neihulizumab in patients with moderate to severe active ulcerative colitis and who has failed or are intolerant to anti-TNFα and/or anti-integrin therapy. A minimum of 30 patients and a maximum of 40 will be recruited in 1 dosing group. For efficacy evaluation, the primary endpoint is the proportion of patients with clinical response, defined as ≥ 3- point reduction in MCS, a 30% or greater decrease from the baseline score, and with a 1-point or greater decrease of the rectal bleeding subscore or an absolute rectal bleeding score of 0 or 1 at Week 12. Safety assessments will consist of evaluating physical examination, vital signs (blood pressure, heart rate, respiratory rate, body temperature and oxygen saturation), safety laboratory tests, adverse events and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent;
2. Age 18-75 years;
3. Diagnosis of UC ≥ 12 weeks prior to screening by full colonoscopy (i.e., ≥ 12 weeks after first diagnosis by a physician according to American College of Gastroenterology guidelines);
4. Moderate-to-severe active UC, at time of screening, defined as:

   1. Mayo Clinic Score (MCS) of 6 points or higher, AND
   2. a centrally read MCS endoscopic subscore of grade 2 or higher, AND
   3. MCS rectal bleeding subscore of 1 point or higher, AND
   4. disease extending 15 cm or more from the anal verge;
5. Stable doses of concomitant medications, including :

   1. Stable oral corticosteroids (i.e., ≤ 20 mg/day of prednisone, ≤ 9 mg/day of budesonide) ≥ 2 weeks before D1 dosing; Taper of oral corticosteroids per Investigator's discretion during the study is allowed;
   2. Stable oral 5-amyinosalicylic acid dose ≥ 2 weeks before D1 dosing;
   3. Stable immunosuppressant including azathioprine, mercaptopurine, or methotrexate ≥ 8 weeks before D1 dosing. Patients taking methotrexate also are advised to take folic acid 1 mg/day or equivalent if there is no contraindication;
   4. Stable doses of probiotics ≥ 2 weeks before D1 dosing;
   5. Stable anti-diarrheas ≥ 2 weeks before D1 dosing;
6. Patients must have previously received anti-tumor necrosis factor alpha (anti- TNF alpha and/or anti-integrin therapy for UC and demonstrated an inadequate response, loss of response, or intolerance, and must have discontinued therapy ≥ 8 weeks before D1 dosing;
7. Patients previously treated with cyclosporine or tacrolimus must have discontinued therapy ≥ 4 weeks before D1 dosing;
8. Topical corticosteroids and topical 5-amyinosalicylic acid preparations must have been withdrawn ≥ 2 weeks before D1 dosing;
9. Nonsteroidal anti-inflammatory drugs (NSAIDs) must have been discontinued ≥ 4 weeks before D1 dosing;
10. Tofacitinib or other Janus kinase (JAK) inhibitors must have been discontinued ≥ 2 weeks before D1 dosing;
11. Patients previously treated with tube feeding, defined formula diets, or parenteral alimentation/nutrition must have discontinued treatment 3 weeks before D1 dosing;
12. Females with reproductive potential must have a negative pregnancy test result before enrollment. Men and women with reproductive potential have to be willing to use a highly effective method of contraception from study start to ≥ 3 months after the final dose of the study drug. A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year).

Exclusion Criteria:

GI related exclusion criteria:

1. Indeterminate colitis (Inflammatory bowel disease unclassified, IBD-U) or suspected Crohn's disease
2. Any history of colectomy
3. Presence of an ileostomy or colostomy
4. A history or evidence of colonic mucosal dysplasia
5. Short gut syndrome

   General health related exclusion criteria:
6. Pregnant or lactating
7. Inability to comply with study protocol in the opinion of the investigator
8. History of dysplasia or malignancy in recent 5 years, except completely excised basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
9. Cirrhosis or active alcohol abuse per the judgement of investigator
10. Poorly controlled diabetes (HbA1c > 8.0%)
11. Significant screening ECG abnormalities, including evidence of acute myocardial infarction, complete left bundle branch block, second-degree heart block, or complete heart block
12. Impaired renal function (calculated creatinine clearance < 60 mL/min)
13. Impaired hepatic function in the absence of diagnosis of primary sclerosing cholangitis, serum transaminase > 2.5x Upper Limit Normal (ULN), alkaline phosphatase > 2.5x ULN, or increased total bilirubin judged by the investigator to be clinically significant, or a diagnosis of primary sclerosing cholangitis, serum transaminases > 3x ULN, alkaline phosphatase > 3x ULN, or total bilirubin > 2.5x ULN judged by the investigator to be clinically significant
14. Moderate to severe anemia (Hb < 8g/dL)
15. Thrombocytopenia (platelet count < 75,000/uL)
16. Evidence of current or previous clinically significant disease, medical condition or finding in the medical examination that in the opinion of the investigator, would compromise the safety of the patient or quality of the data
17. Requiring parenteral corticosteroid treatment.
18. Received any investigational product within 1 year.
19. History of drug abuse according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria within 12 months prior to screening or positive drug screening tests.

    Infection related exclusion criteria:
20. Human immune deficiency virus (HIV) infection or known HIV-related malignancy.
21. Acute or chronic hepatitis B or C, or carrier status. Patients with anti-HBc Ab but with undetectable anti-HBs Ab should also be excluded.
22. Positive IgM antibody titers in the presence of negative IgG titers to Epstein-Barr virus
23. Positive stool test for ova or parasites, positive stool culture for pathogens, or positive stool toxin assay for Clostridium difficile at screening. Patients with the positive stool toxin assay for C. difficile at screening could be rescreened if they are being treated for C. difficile and a repeat stool toxin assay at least 4 weeks after the completion of treatment is negative with no evidence of recurrence.
24. Intestinal mucosa biopsy positive for cytomegalovirus (CMV) at screening.
25. Positive screening test for latent Mycobacterium tuberculosis (TB) infection. Patients with a history of latent TB infection who received an appropriate and documented course of therapy can be included if the screening examination and a chest x-ray performed ≤ 3 months before screening revealed no evidence of current active infection. If a Quantiferon TB test is indeterminate, the test should be repeated, and if the result is again indeterminate, such patient should be excluded.
26. History of any opportunistic infection ≤ 12 weeks before D1 dosing.
27. Any current or recent (≤ 4 weeks before D1 dosing) symptoms/signs of infection.
28. Received oral antibiotics ≤ 4 weeks before D1 dosing or intravenous antibiotics ≤ 8 weeks before D1 dosing.
29. Received a live attenuated vaccine ≤ 4 weeks before D1 dosing.
30. Neutropenia (absolute neutrophil count < 1,500/uL).
31. Lymphocytopenia (absolute lymphocyte count < 500 /uL).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yao Lin, MD, PhD, Study Director — AltruBio Inc.; David T Rubin, MD, Principal Investigator — University of Chicago
Locations (12):
- United States (11):
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Stomach Doctor - Surinder Saini, MD - Fountain Valley, Newport Beach, California
  - Wellness Clinical Research (WCR), Hialeah, Florida
  - Wellness Clinical Research (WCR), Lake Wales, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Capitol Research, Rockville, Maryland
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Baylor College of Medicine, Houston, Texas
  - University of Washington Medical Center (UWMC) - Digestive Disease Center, Seattle, Washington
- Wellness Clinical Research (WCR), Vega Baja, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 12 centers locate in North America and Puerto Rico from May 2018 to June 2020. It was a 24 weeks open label, single arm, multiple dose proof of principle study.
Groups:
- ALTB-168 in Patients With Refractory Ulcerative Colitis: Amendment 1~3: 9 mg/kg; total of 8 doses of ALTB-168. Amendment 4: 9 mg/kg; total of 10 doses of ALTB-168.
Period: Overall Study
Arm/Group | ALTB-168 in Patients With Refractory Ulcerative Colitis
Started | 24
Number of Participants Who Received 8 Doses of ALTB-168 | 10
Number of Participants Who Received 10 Doses of ALTB-168 | 14
Completed | 11
Not Completed | 13
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 1
Not completed — disease relapse | 1

BASELINE CHARACTERISTICS:
Population: Safety population /The mITT set was defined as all patients who were enrolled and who received at least one dose of ALTB-168 treatment.
Arm/Group | ALTB-168
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — Population: Total enrolled number of participants is 24. 10 participants were enrolled under Amendment 1-3 14 participants were enrolled under Amendment 4
  Participants
    Enrolled Under Amendment 1-3: number analyzed (Participants) | 10
    Enrolled Under Amendment 1-3: <=18 years | 0
    Enrolled Under Amendment 1-3: Between 18 and 65 years | 9
    Enrolled Under Amendment 1-3: >=65 years | 1
    Enrolled Under Amendment 4: number analyzed (Participants) | 14
    Enrolled Under Amendment 4: <=18 years | 0
    Enrolled Under Amendment 4: Between 18 and 65 years | 14
    Enrolled Under Amendment 4: >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] — Population: 10 subjects were enrolled under Amendment 1-3 and 14 subjects under Amendment 4.
  years
    Amendment 1-3: number analyzed (Participants) | 10
    Amendment 1-3 | 37 [21 to 65]
    Amendment 4: number analyzed (Participants) | 14
    Amendment 4 | 35.5 [22 to 61]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Row population does not differ from the Overall population. Altogether 24 participants were enrolled to the study. Out of them 10 were enrolled under protocol Amendments 1-3 and 14 under the Amendment 14.
  Participants
    Enrolled under Amendment 1~3: number analyzed (Participants) | 10
    Enrolled under Amendment 1~3: Female | 6
    Enrolled under Amendment 1~3: Male | 4
    Enrolled under Amendment 4: number analyzed (Participants) | 14
    Enrolled under Amendment 4: Female | 7
    Enrolled under Amendment 4: Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 7
  Ethnicity: Not Hispanic or Latino | 15
  Ethnicity: Not reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients With Clinical Response at Week 12
Description: The clinical response is defined as a ≥ 3-point reduction in Mayo Clinic Score, a 30% or greater decrease from the baseline score, and with a 1-point or greater decrease of the rectal bleeding subscore or an absolute rectal bleeding score of 0 or 1,
  The colonic site with maximum inflammation was determined by Mayo endoscopic subscore (MES) defined as follows: normal (0 points); erythema, decreased vascular pattern, mild friability (1 point); absent vascular pattern, friability, erosions (2 points); and spontaneous bleeding or ulceration (3 points).
  Lower score means disease improvement.
Time Frame: week 12
Population: The full analysis set includes all participants who received at least 1 dose of study drug. The response rates were calculated using non-responder imputation, where participants with a missing scores at week 12 were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of total number of patients
Groups:
- Pilot Study (Amendment 1~3: 9 mg/kg; Total 8 Doses): 10 participants enrolled under protocol Amendments 1-3 received total of 8 doses of ALTB-168
- Main Study (Amendment 4: 9 mg/kg; Total 10 Doses): 14 participants enrolled under Amendment 4 received total of 10 doses of ALTB-168
Arm/Group | Pilot Study (Amendment 1~3: 9 mg/kg; Total 8 Doses) | Main Study (Amendment 4: 9 mg/kg; Total 10 Doses)
Number analyzed (Participants) | 9 | 14
percentage of total number of patients | 22.2 [2.8 to 60] | 50 [23 to 77]

2. Secondary Outcome: The Proportion of Patients With Clinical Response (mITT)
Description: The proportion of patients with clinical response defined as a ≥2-point decrease in partial MCS (pMCS), and with a 1 point or greater decrease of the rectal bleeding subscale or an absolute rectal bleeding score of 0 or 1.
  The colonic site with maximum inflammation was determined by Mayo endoscopic subscore (MES) defined as follows: normal (0 points); erythema, decreased vascular pattern, mild friability (1 point); absent vascular pattern, friability, erosions (2 points); and spontaneous bleeding or ulceration (3 points).
  Lower score means disease improvement.
Time Frame: weeks 6,16, 20 and 26
Population: The full analysis set includes all participants who received at least 1 dose of study drug. Response rates were calculated using non-responder imputation, where participants with a missing information were counted as non-responders. 23 participants are included in the study analysis. 9 participants from the pilot study (protocol Amendments 1-3) and 14 participants from the main study (protocol Amendment 4).
Measure: Number (95% Confidence Interval); unit: percentage of total number of patients
Groups:
- Pilot Study (Amendment 1~3: 9 mg/kg; Total 8 Doses): 10 participants were enrolled under Amendments 1-3 of the study protocol
- Main Study (Amendment 4: 9 mg/kg; Total 10 Doses): 14 participants were enrolled under Amendment 4 of the study protocol
Arm/Group | Pilot Study (Amendment 1~3: 9 mg/kg; Total 8 Doses) | Main Study (Amendment 4: 9 mg/kg; Total 10 Doses)
Number analyzed (Participants) | 9 | 14
percentage of total number of patients
  Clinical Response at week 6 | 33.3 [7.5 to 70.1] | 57.1 [28.9 to 82.3]
  Clinical Response at week 16 | 0 [0 to 0] | 64.3 [35.1 to 87.2]
  Clinical Response at week 20 | 11.1 [0.3 to 48.2] | 64.3 [35.1 to 87.2]
  Clinical Response at week 26 | 11.1 [0.3 to 48.2] | 35.7 [12.8 to 64.9]

3. Secondary Outcome: The Proportion of Patients With Clinical Remission
Description: The number of patients with clinical remission, defined as MCS of 2 or lower (or pMCS of 1 or lower) and no subscore higher than 1.
  The colonic site with maximum inflammation was determined by Mayo endoscopic subscore (MES) defined as follows: normal (0 points); erythema, decreased vascular pattern, mild friability (1 point); absent vascular pattern, friability, erosions (2 points); and spontaneous bleeding or ulceration (3 points).
  Lower score means disease improvement.
Time Frame: weeks 6,16, 20 and 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of total number of patients
Groups:
- Amendment 1~3: 9 mg/kg; Total 8 Doses: Amendment 1~3: 9 mg/kg; total 8 doses of ALTB-168
- Amendment 4: 9 mg/kg; Total 10 Doses: Amendment 4: 9 mg/kg; total 10 doses of ALTB-168
Arm/Group | Amendment 1~3: 9 mg/kg; Total 8 Doses | Amendment 4: 9 mg/kg; Total 10 Doses
Number analyzed (Participants) | 9 | 14
percentage of total number of patients
  Clinical response at week 6 | 11.1 [0.3 to 48.2] | 35.7 [12.8 to 64.9]
  Clinical response at week 16 | 0 [0 to 0] | 35.7 [12.8 to 64.9]
  Clinical response at week 20 | 0 [0 to 0] | 35.7 [12.8 to 64.9]
  Clinical response at week 26 | 11.1 [0.3 to 48.2] | 21.4 [4.7 to 50.8]

4. Secondary Outcome: Flexible Sigmoidoscopy Subscore Changes From Baseline
Description: The mean (SD) observed flexible sigmoidoscopy subscore change from baseline (CFB).
  Baseline is defined as the last available assessment prior to the first administration of the study drug. The sigmoidoscopic improvement is defined as any decrease in Mayo Clinic Score (MCS) endoscopic subscore, at Weeks 12 and 26. MCS range is 1-3.
  The colonic site with maximum inflammation was determined by Mayo endoscopic subscore (MES) defined as follows: normal (0 points); erythema, decreased vascular pattern, mild friability (1 point); absent vascular pattern, friability, erosions (2 points); and spontaneous bleeding or ulceration (3 points).
  Lower score means disease improvement.
Time Frame: Baseline, week 12- and week 26 after the first treatment
Population: Study participants who entered the study under amendment 1-3 (n=9) and participans who entered the study under amendment 4 (n=14) have been inlcuded in this analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amendment 1~3: 9 mg/kg; Total 8 Doses | Amendment 4: 9 mg/kg; Total 10 Doses
Number analyzed (Participants) | 9 | 14
score on a scale
  Flexible Sigmoidoscopy Score at Baseline | 2.7 (0.5) | 2.6 (0.5)
  Flexible Sigmoidoscopy Score at week 12 CFB | -0.7 (1.03) | -0.6 (1.0)
  Flexible Sigmoidoscopy Score at week 26 CFB | 0 (0) | -0.6 (1.27)

5. Secondary Outcome: The Number of Patients With Mucosal Healing
Description: The mucosal healing is defined as an absolute subscore for endoscopy of 0 or 1 The colonic site with maximum inflammation was determined by Mayo endoscopic subscore (MES) defined as follows: normal (0 points); erythema, decreased vascular pattern, mild friability (1 point); absent vascular pattern, friability, erosions (2 points); and spontaneous bleeding or ulceration (3 points).
  Lower score means disease improvement.
Time Frame: at 12- and 26-week after the first treatment
Population: Study participants who received at least one dose of ALTB-168. Missing data imputed as non-responders (i.e. Amd 1-3: Week 12 - 3 missing; Week 26 - 8 missing; and Amd 4: Week 12 - 2 missing; Week 26 - 7 missing).
Measure: Number; unit: participants
Arm/Group | Amendment 1~3: 9 mg/kg; Total 8 Doses | Amendment 4: 9 mg/kg; Total 10 Doses
Number analyzed (Participants) | 9 | 14
participants
  Week 12 | 2 | 4
  Week 26 | 0 | 3

6. Secondary Outcome: Change of Histological Activity Grade From Baseline Using the Geboes System
Description: The number of patients with histological activity Geboes Score ≤ 3.1 (worst of both rectum and sigmoid colon).
  The original Geboes grade system is from Grade 0 to Grade 5.
  The following are the grades:
  Grade 0: Architectural changes Grade 1: Chronic inflammatory infiltrate Grade 2A: Eosinophils in lamina propria Grade 2B: Neutrophils in lamina propria Grade 3: Neutrophils in epithelium Grade 4:Crypt destruction Grade 5: Erosions and ulcerations
Time Frame: at 12- and 26-week after the first treatment
Population: Study participants who received at least one dose of ALTB-168
Measure: Number; unit: participants
Arm/Group | Amendment 1~3: 9 mg/kg; Total 8 Doses | Amendment 4: 9 mg/kg; Total 10 Doses
Number analyzed (Participants) | 9 | 14
participants
  Week 12: number analyzed (Participants) | 9 | 12
  Week 12 | 0 | 2
  Week 26: number analyzed (Participants) | 9 | 12
  Week 26 | 1 | 4

7. Secondary Outcome: The Number of Patients With Histological Healing
Description: The histological healing is defined as histological grade = 0
Time Frame: at 12- and 26-week after the first treatment
Population: Study participants who received at least one dose of ALTB-168. Missing data imputed as non-responders (i.e. Amd 1-3: Week 12 - 4 missing; Week 26 - 8 missing; and Amd 4: Week 12 - 2 missing; Week 26 - 7 missing).
Measure: Count of Participants; unit: Participants
Arm/Group | Amendment 1~3: 9 mg/kg; Total 8 Doses | Amendment 4: 9 mg/kg; Total 10 Doses
Number analyzed (Participants) | 9 | 14
Participants
  Week 12 | 0 | 0
  Week 26 | 0 | 0

8. Secondary Outcome: Change of Inflammatory Bowel Disease Questionnaire (IBDQ) Score From Baseline
Description: Number of Participants with a Clinically Significant Difference in the Inflammatory Bowel Disease Questionnaire (IBDQ) Score From Baseline, to Week 12 and Week 26.
  The IBDQ is a questionnaire used for an assessment of Health Related Quality of Life (HRQoL) in patients with the Inflammatory Bowel Disease (IBD). The IBDQ has a possible score range of 32 (minimum) to 224 (maximum), where a higher score indicates better HRQoL. A difference of 16 points from Baseline Assessment (Baseline Score) to Week 12, and Baseline Assessment (Baseline Score) to Week 26, is considered clinically significant. The outcome measure is assessed by comparing each patient's change in individual IBDQ score from Baseline to Week 12, and from Baseline to Week 26. Patients who achieved the 16 point difference (improvement of the IBDQ score from the baseline indicating the Clinically Significant Difference) are included as responders to the treatment.
Time Frame: at 12- and 26-week after the first treatment
Population: Study participants who received at least one dose of ALTB-168. Missing data imputed as non-responders (i.e. Amd 1-3: Week 12 - 3 missing; Week 26 - 8 missing; and Amd 4: Week 12 - 0 missing; Week 26 - 6 missing).
Measure: Number; unit: participants
Arm/Group | Amendment 1~3: 9 mg/kg; Total 8 Doses | Amendment 4: 9 mg/kg; Total 10 Doses
Number analyzed (Participants) | 9 | 14
participants
  Week 12 | 2 | 9
  Week 26 | 1 | 7

9. Secondary Outcome: The Number of Patients With Inflammatory IBDQ Response
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) has a possible score range of 32 (minimum) to 224 (maximum), where a higher score indicates better Health Related Quality of Life (HRQoL). A difference of 16 points from Baseline to Week 12 and Baseline to Week 26, is considered clinically significant. The outcome measure will be assessed by comparing each patient's change in individual IBDQ score from Baseline to Week 12, and from Baseline to Week 26, to assess whether a response was seen.
Time Frame: at 12- and 26-week after the first treatment
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Amendment 1~3: 9 mg/kg; Total 8 Doses | Amendment 4: 9 mg/kg; Total 10 Doses
Number analyzed (Participants) | 9 | 14
participants
  Week 12 | 2 | 9
  Week 26 | 1 | 7

10. Other Pre Specified Outcome: CRP Changes From Baseline (CFB) (Exploratory)
Description: Change in biomarkers of CRP (C-reactive protein). C-reactive protein (CRP) is a biomarker produced by your liver in response to inflammation. Normal CRP value is below 1 mg/L.
  1-3 mg/L is in the "yellow zone", indicating some inflammation >3 mg/L is in the "red zone", meaning there is significant inflammation
Time Frame: Am 4, Weeks 4, 9, 12, 16, 20, 26; Am 1-3 weeks 4,8,12,16,20, 26
Population: Study participants who received at least one dose of ALTB-168
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Amendment 1~3: 9 mg/kg; Total 8 Doses | Amendment 4: 9 mg/kg; Total 10 Doses
Number analyzed (Participants) | 9 | 14
mg/L
  Baseline | 4.3 (5.32) | 11.29 (20.555)
  Week 4: number analyzed (Participants) | 8 | 14
  Week 4 | 6.5 (17.30) | -1.93 (14.403)
  Am 4 Week 9, Am 1-3 Week 8: number analyzed (Participants) | 6 | 13
  Am 4 Week 9, Am 1-3 Week 8 | 6.2 (10.65) | -0.42 (18.821)
  Week 12: number analyzed (Participants) | 2 | 13
  Week 12 | 6.0 (8.49) | 0.12 (15.605)
  Week 16: number analyzed (Participants) | 1 | 10
  Week 16 | NA (NA) — Only 1 participant | -0.65 (13.450)
  Week 20: number analyzed (Participants) | 1 | 9
  Week 20 | NA (NA) — Only 1 participant | -2.94 (14.161)
  Week 26: number analyzed (Participants) | 1 | 6
  Week 26 | NA (NA) — Only 1 participant | -0.42 (4.079)

11. Other Pre Specified Outcome: Changes in Fecal Calprotectin (CFB) - Exploratory Biomarker
Description: Faecal calprotectin changes from the baseline at Week 4, 9, 12, 16, 20, and 26 were measured. Baseline is defined as the last available assessment prior to the first administration of the study drug.
  Faecal calprotectin is measured as mcg/g, so the results come back as a numeric value. A level under 50 is considered to be 'normal'. A level between 50 and 100, coupled with digestive symptoms, means IBS is likely. Lower level means improvement.
Time Frame: Am 4, Weeks 4, 9, 12, 16, 20, 26; Am 1-3 weeks 4,8,12,16,20, 26
Population: Study participants who received at least one dose of ALTB-168
Measure: Mean (Standard Deviation); unit: mcg/g
Arm/Group | Amendment 1~3: 9 mg/kg; Total 8 Doses | Amendment 4: 9 mg/kg; Total 10 Doses
Number analyzed (Participants) | 9 | 14
mcg/g
  Baseline | 682.80 (548.153) | 1283.49 (758.019)
  Week 4 (CFB): number analyzed (Participants) | 8 | 12
  Week 4 (CFB) | 113.89 (753.179) | -203.30 (704.559)
  Week 9 (Am 4, week 8 Am 1-3): number analyzed (Participants) | 6 | 13
  Week 9 (Am 4, week 8 Am 1-3) | 223.17 (605.971) | -384.47 (662.420)
  Week 12: number analyzed (Participants) | 2 | 13
  Week 12 | 923.00 (997.162) | -584.17 (847.809)
  Week 16: number analyzed (Participants) | 1 | 9
  Week 16 | NA (NA) — Only 1 participant | -155.01 (1142.984)
  Week 20: number analyzed (Participants) | 1 | 8
  Week 20 | NA (NA) — Only 1 participant | -29.46 (477.150)
  Week 26: number analyzed (Participants) | 1 | 5
  Week 26 | NA (NA) — Only 1 participant | -780.30 (633.292)

ADVERSE EVENTS:
Time Frame: 26 weeks
Groups:
- ALTB-168 9mg/kg (Amendment 1-3): Amendments 1-3: A total of 8 doses of ALTB-168 at 9 mg/kg
- ALTB-168 9mg/kg (Amendment 4): Amendment 4: A total of 10 doses of ALTB-168 at 9 mg/kg
Arm/Group | ALTB-168 9mg/kg (Amendment 1-3) | ALTB-168 9mg/kg (Amendment 4)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/14
Other Adverse Events (participants affected / at risk) | 9/10 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALTB-168 9mg/kg (Amendment 1-3) (N=10) | ALTB-168 9mg/kg (Amendment 4) (N=14)
Ulcerative Colitis Flare (Gastrointestinal disorders) | 1 (1) | 0 — Participant ID AE Term Date of onset AE Outcome Relatedness to IP 1010003 Ulcerative Colitis flare 05AUG2018 Resolved Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALTB-168 9mg/kg (Amendment 1-3) (N=10) | ALTB-168 9mg/kg (Amendment 4) (N=14)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 1
Headache (Nervous system disorders) | 5 (5) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Confusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Fecal Calprotectin Increased (Investigations) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Palate Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear Swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Body Tinea (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT03298022/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT03298022/SAP_001.pdf
  • Informed Consent Form (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT03298022/ICF_002.pdf